CLINICAL TRIAL: NCT00464503
Title: The Effect of Statins on the Urinary Proteome
Brief Title: Statins and the Urinary Proteome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: STAT-AZ-01
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Statin Induced Proteinuria
Keywords: statins; proteinuria; proteomic analysis; healthy volunteers
MeSH Terms: conditions — Proteinuria | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rosuvastatin-Crestor
Drug: Pravastatin-Pravasine

SUMMARY:
This study aims to investigate whether statines (rosuva- and pravastatin) induce tubular proteinuria.

DETAILED DESCRIPTION:
The proximal tubular cells of the kidney are responsible for reabsorption of proteins from the tubular lumen. In a study using Opossum kidney (OK) cells, receptor-mediated protein endocytosis was reduced by statins, inhibitors of 3-hydroxy-3-methylglutaryl CoA (HMG-CoA) reductase, which are widely used for therapeutic reduction of plasma cholesterol levels (1). In a subsequent in vitro study protein endocytosis in human mixed proximal/distal kidney tubular cells was investigated in the presence and absence of statins to explore the possible clinical relevance of the observations in OK cells (2). The uptake of FITC-labeled albumin in these cultures occurred selectively into proximal tubular cells while it was absent in distal tubular/collecting duct cells. Three statins (simvastatin, pravastatin, and rosuvastatin) significantly inhibited the uptake of protein in a concentration-dependent way. This inhibitory effect of statins could be prevented by the co-addition of mevalonate, the product of HMG-CoA reductase. This effect was not the result of a statin-induced cytotoxicity since cell-viability was unaffected.

These data suggest that statins have the potential to inhibit albumin uptake by the human proximal nephron as a result of inhibition of HMG-CoA reductase in the proximal tubule cells. A reduced prenylation of some proteins critically involved in endocytosis has been put forward as the underlying mechanism.

Knowing these data it has been suggested that the occurrence of proteinuria in some patients treated with high statin doses is the result of a reduced tubular reabsorption/endocytosis of normally filtered proteins. To further explore the clinical relevance of such a mechanism, the composition of the urinary proteome under statin treatment will be investigated in normal healthy volunteers by two-dimensional gel electrophoresis based proteomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male, age range: 25 - 65 years
* Non-smoker
* Proteinuria: < 60 mg/24 hours
* Dipstick negative hematuria
* Bloodpressure: < 135 mm systolic, < 85 mm dyastolic
* Waist circumference: < 94 cm

Exclusion Criteria:

* Treatment with lipid-lowering drugs <1 year prior to the study
* Known history of diabetes or fasting glucose level: < 110 mg/dl
* Anti-hypertensive medication
* Life-expectancy < 1 year
* Pharmacological treatment with inotropes
* Acute or chronic inflammatory process, use if anti-inflammatory drugs or immunosuppression
* Clinically active malignant disease
* Administration of any investigational drug within 30 days preceding study start and during the study
* Known intolerance to rosuvastatin or other statins
* Acute or chronic liver disease or ALAT>2.0 x upper limit of normal (ULN) at enrolment visit.
* Chronic muscle disease such as dermatomyositis or polymyositis or unexplained creatinine kinase (CK) above 3 x ULN at enrolment.
* Uncontrolled hypothyroidism as indicated by a thyroid stimulating hormone (TSH) > 2 x ULN at enrolment.
* Renal insufficiency: creatinine > 2.0mg/dl
* Known or suspect alcohol or drug abuse.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The urinary protein pattern observed by difference gel electrophoresis based proteomics analysis in healthy subjects before and after the administration of rosuvastatin (Crestor®).

SECONDARY OUTCOMES:
The urinary protein pattern observed by difference gel electrophoresis based proteomics analysis in healthy subjects before and during the administration of pravastatin (Pravasine®).
The urinary protein pattern observed by difference gel electrophoresis based proteomics analysis in healthy subjects during the administration of rosuvastatin (Crestor®) vs pravastatin (Pravasine®).
The urinary protein pattern observed by difference gel electrophoresis based proteomics analysis in healthy subjects during the administration of rosuvastatin (Crestor®) or pravastatin (Pravasine®) and after wash-out of these compounds.
The urinary albumin and retinol binding protein concentration before in healthy subjects, during and after administration of rosuvastatin (Crestor®) or pravastatin (Pravasine®).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick C D'Haese, Prof, Study Director — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Antwerp, Antwerp, Belgium